CLINICAL TRIAL: NCT03778957
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter Study of Transarterial Chemoembolization (TACE) in Combination With Either Durvalumab Monotherapy or Durvalumab Plus Bevacizumab Therapy in Patients With Locoregional Hepatocellular Carcinoma (EMERALD-1)
Brief Title: A Global Study to Evaluate Transarterial Chemoembolization (TACE) in Combination With Durvalumab and Bevacizumab Therapy in Patients With Locoregional Hepatocellular Carcinoma
Acronym: EMERALD-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D933GC00001; 2023-509053-32-00 (Registry Identifier: CTIS (EU)); 2018-002134-20 (EudraCT Number)
Record Dates: First submitted 2018-11-28; First posted 2018-12-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; TACE; Durvalumab; Bevacizumab; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — durvalumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Transarterial Chemoembolization (TACE) in combination with Durvalumab
  Interventions: Drug: Durvalumab; Other: Placebo; Procedure: Transarterial Chemoembolization (TACE)
- Arm B (Experimental): Transarterial Chemoembolization (TACE) in combination with Durvalumab and Bevacizumab
  Interventions: Drug: Durvalumab; Drug: Bevacizumab; Procedure: Transarterial Chemoembolization (TACE)
- Arm C (Placebo Comparator): Transarterial Chemoembolization (TACE) in combination with Placebos
  Interventions: Other: Placebo; Procedure: Transarterial Chemoembolization (TACE)

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (intravenous)
  Other Names: MEDI4736
  Arms: Arm A; Arm B
Drug: Bevacizumab — Bevacizumab IV (intravenous)
  Other Names: AVASTIN
  Arms: Arm B
Other: Placebo — Saline solution for Durvalumab and/or Bevacizumab masking (IV intravenous)
  Arms: Arm A; Arm C
Procedure: Transarterial Chemoembolization (TACE) — TACE (chemo and embolic agent injection into the hepatic artery)

SUMMARY:
A global study to evaluate transarterial chemoembolization (TACE) in combination with durvalumab and bevacizumab therapy in patients with locoregional hepatocellular carcinoma

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter, global Phase III study to determine the efficacy and safety of transarterial chemoembolization (TACE) treatment in combination with durvalumab monotherapy or TACE given with durvalumab plus bevacizumab therapy compared to TACE therapy alone in patients with locoregional hepatocellular carcinoma not amenable to curative therapy

ELIGIBILITY:
Key Inclusion Criteria:

* No evidence of extrahepatic disease
* Disease not amenable to curative surgery or transplantation or curative ablation but disease amenable to TACE
* Child-Pugh score class A to B7 and Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
* Measurable disease by Modified Response Criteria in Solid Tumors (mRECIST) criteria
* Adequate organ and marrow function

Key Exclusion Criteria

* Any history of nephrotic or nephritic syndrome
* Clinically significant cardiovascular disease or history of arterioembolic event including a stroke or myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack within 6 months prior to randomization
* Any prior or current evidence of coagulopathy or bleeding diathesis or patients who had any kind of surgery in the past 28 days (biopsies are exempt from this exclusion)
* History of abdominal fistula or GI perforation, non healed gastric ulcer that is refractory to treatment, or active GI bleeding within 6 months prior to enrollment
* Patients with Vp3 and Vp4 portal vein thrombosis on baseline imaging are excluded

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) for Arm B vs Arm C | Approximately 5 years
  PFS per Blinded Independent Central Review (BICR) assessment will be defined as the time from the date of randomization until the date of first objective disease progression or death

SECONDARY OUTCOMES:
Progression Free Survival (PFS) for Arm A vs Arm C | Approximately 5 years
  PFS per Blinded Independent Central Review (BICR) assessment will be defined as the time from the date of randomization until the date of first objective disease progression or death
Overall Survival (OS) | Approximately 5 years
  OS is defined as the time from the date of randomization until death due to any cause
Health status/quality of life measured by European Organization for Research and Treatment of Cancer (EORTC) 30-item core quality of life questionnaire (QLQ-C30) | Approximately 5 years
  Collection of patient reported outcome (PRO) measures to assess time to deterioration in global health status/quality of life (QoL), functioning (physical) and symptoms
Disease-related symptoms measured by European Organization for Research and Treatment of Cancer (EORTC) 18-item hepatocellular cancer health-related quality of life questionnaire (QLQ-HCC18) | Approximately 5 years
  Collection of patient reported outcome (PRO) measures to assess time to deterioration in symptoms

OTHER OUTCOMES:
Safety of Durvalumab and Bevacizumab as evaluated by summary of adverse events by treatment arm and CTCAE grade | Approximately 5 years
Immunogenicity of Durvalumab and Bevacizumab as measured by presence of anti-drug antibodies (ADAs) | Approximately 5 years
Pharmacokinetics (PK) of Durvalumab and Bevacizumab as determined by peak serum concentrations | Approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Sangro, MD, Principal Investigator — Clinica Universidad de Navarra; Riccardo Lencioni, MD FSIR EBIR, Principal Investigator — University of Pisa / Miami Cancer Institute
Locations (138):
- United States (22):
  - Research Site, Costa Mesa, California
  - Research Site, La Jolla, California
  - Research Site, Orange, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Shreveport, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Stony Brook, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin
- Australia (7):
  - Research Site, Benowa
  - Research Site, Box Hill
  - Research Site, Camperdown
  - Research Site, Clayton
  - Research Site, Herston
  - Research Site, Liverpool
  - Research Site, Melbourne
- Brazil (8):
  - Research Site, Barretos
  - Research Site, Florianópolis
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santa Maria
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Vitória
- Canada (3):
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (21):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nantong
  - Research Site, Neijiang
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
  - Research Site, Zhuhai
- France (9):
  - Research Site, Bobigny
  - Research Site, Clichy
  - Research Site, Grenoble
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- India (11):
  - Research Site, Bangalore
  - Research Site, Bengaluru
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, Mumbai
  - Research Site, Nashik
  - Research Site, Pune
  - Research Site, Surat
  - Research Site, Vijayawada
  - Research Site, Visakhapatnam
- Italy (4):
  - Research Site, Arezzo
  - Research Site, Brescia
  - Research Site, Milan
  - Research Site, Pisa
- Japan (15):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kurume-shi
  - Research Site, Musashino-shi
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Shiwa-gun
  - Research Site, Tsu
  - Research Site, Yokohama
- Mexico (7):
  - Research Site, Alc. Cuauhtémoc
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Mérida
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Tuxtla Gutiérrez
- Russia (7):
  - Research Site, Barnaul
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Yekaterinburg
- Research Site, Singapore, Singapore
- South Korea (4):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (4):
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, San Sebastián(Guipuzcoa)
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, Liou Ying Township
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Phisanulok
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Sangro B, Kudo M, Erinjeri JP, Qin S, Ren Z, Chan SL, Arai Y, Heo J, Mai A, Escobar J, Lopez Chuken YA, Yoon JH, Tak WY, Breder VV, Suttichaimongkol T, Bouattour M, Lin SM, Peron JM, Nguyen QT, Yan L, Chiu CF, Santos FA, Veluvolu A, Thungappa SC, Matos M, Zotkiewicz M, Udoye SI, Kurland JF, Cohen GJ, Lencioni R; EMERALD-1 Investigators. Durvalumab with or without bevacizumab with transarterial chemoembolisation in hepatocellular carcinoma (EMERALD-1): a multiregional, randomised, double-blind, placebo-controlled, phase 3 study. Lancet. 2025 Jan 18;405(10474):216-232. doi: 10.1016/S0140-6736(24)02551-0. Epub 2025 Jan 8. PMID 39798579
- [Derived] Kloeckner R, Galle PR, Bruix J. Local and Regional Therapies for Hepatocellular Carcinoma. Hepatology. 2021 Jan;73 Suppl 1:137-149. doi: 10.1002/hep.31424. Epub 2020 Nov 6. No abstract available. PMID 32557715